CLINICAL TRIAL: NCT02394587
Title: A Mindfulness-based Intervention For Pain Catastrophizing In Sickle Cell Disease
Brief Title: MBSR for Pain Catastrophizing in SCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00052848; F31NR014954-01 (NIH)
Record Dates: First submitted 2015-02-09; First posted 2015-03-20 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-04

CONDITIONS: Anemia, Sickle Cell
Keywords: mindfulness; MBSR; SCD; experimental
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-Based Stress Reduction (Experimental): Subjects assigned to the experimental group will participate in a MBSR foundation program, which includes weekly telephonic, group-based, 60-minute MBSR sessions for 6 weeks. The foundation program will introduce subjects to the concept of mindfulness with each week focusing on a different facet. Modeled after Kabat-Zinn's original program, breath awareness (focus on breath and observing thoughts without fighting or following them), body scan (promoting mindfulness of sensations in different parts of body), walking meditation (walking as form of meditation), loving kindness (projection of friendliness and kindness towards oneself and others), and choiceness awareness (awareness of all sensations with equal interest) will be taught.
  Interventions: Behavioral: Mindfulness-based Stress Reduction
- Wait-listed control group (Other): Subjects assigned to the wait-listed control group will not receive the MBSR program, but will receive weekly reminders of their study participation, be asked to complete the same questionnaires (per telephone script) once every three weeks, and receive the same financial incentives as the MBSR group. Upon completion of the 6-week session, the wait-list control group will be offered the same MBSR program. At that time, a new series of MBSR sessions will be scheduled and offered to the wait-listed control patients. Subjects who elect to participate in MBSR will receive the same packet of materials and measures received by the intervention group and be asked to complete the measures again at baseline, 1, 3, and 6 weeks.
  Interventions: Behavioral: Mindfulness-based Stress Reduction

INTERVENTIONS:
Behavioral: Mindfulness-based Stress Reduction — A non-pharmacological approach to pain management.

SUMMARY:
Significance: The purpose of this exploratory study is to test the feasibility, accessibility, and effects of a mindfulness-based stress reduction program (MBSR) on reducing pain catastrophizing in persons with sickle cell disease (SCD) and chronic pain. One of the most difficult symptoms for SCD patients to manage is chronic pain. Approximately one-third of SCD patients experience chronic pain, which is associated with pain catastrophizing. Pain catastrophizing is a negative mental state toward pain stimuli and pain experience, and is associated with increased pain severity, pain interference, and lower social functioning, physical functioning, and mental health. There have been no psychobehavioral intervention studies that have attempted to alter the experience of pain catastrophizing in persons with SCD. MBSR is a complementary group-based therapy that emphasizes nonjudgmental awareness of thoughts, feelings, and bodily sensations. With no pharmacological or non-pharmacological treatment for catastrophizing in persons with SCD, MBSR offers a potential solution to this highly significant problem for both SCD patients and providers. This project will be the first randomized controlled trial (RCT) of MBSR to reduce pain catastrophizing, and improve quality of life for SCD patients with chronic pain.

Methods: This study will enroll 60 adult patients with SCD and chronic pain from the Duke Adult Sickle Cell Clinic. Patients will be randomized to a MBSR or wait-listed control group. The MBSR group will complete a 6- week, group-based telephonic MBSR program that is administered by a certified MBSR clinician once a week for 90 minutes. MBSR feasibility, acceptability, and effects on pain catastrophizing will be assessed by questionnaires at baseline, week 1, 3, and 6 in both groups. At the end of week 6, 10 randomly selected MBSR participants will complete semi-scripted telephone interviews to help assess intervention acceptability, and the wait-listed control condition will be offered the same MBSR intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent,
2. Are >age 21,
3. Self-identify (to the PI at baseline assessment) that they are experiencing chronic, non-cancer pain that has persisted on most days for more than 6 months, and adversely affects their function or well-being,
4. are able to speak and read English,
5. Have access to a telephone (or cell phone) in the home for the intervention and individual assessment interviews (data from the SCD clinic indicate 82% of patients have a cell phone),
6. Have access to a CD or mp3 player for homework assignments and daily practice,
7. Are available during the scheduled telephone intervention, and
8. Complete and return the baseline assessment

Exclusion Criteria:

* Patients will be excluded if they report previously studying MBSR, currently receiving mindfulness-based or cognitive behavioral therapies, or being regular practitioners of mindfulness, including yoga.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of MBSR as measured by semi-scripted telephone assessments | 6 weeks
  Acceptability of the intervention will be assessed by semi-scripted telephone or in-person interviews. The semi-scripted interview will focus on MBSR patients' reflections and expectations of the program, the mindfulness skills they found useful and in what ways, the skills they found less useful and or difficult to implement, and on any changes in thoughts or actions that resulted from the application of the MBSR techniques.
Feasibility of MBSR as measured by recruitment, attrition rates, and practice logs | 6 weeks
  Feasibility of the intervention will be assessed by recruitment and attrition rates, number of daily mindfulness logs completed, and average number of weekly minutes of mindfulness practice as recorded in logs. Feasibility data will be obtained for both the intervention and control subjects who elect to receive the intervention after the intervention is complete with the MBSR group. However, data will not be analyzed together because the delay to receiving the intervention would affect the results. Data from the control group will be used to help inform future studies.

SECONDARY OUTCOMES:
Change in Pain Catastrophizing as measured by the Pain Catastrophizing Scale | baseline, week 1, week 3, and week 6
  Descriptive statistics will be used to summarize the pain catastrophizing at week1, 3, and 6, as measured by the Pain Catastrophizing Scale. Trajectory analyses, using a type of mixed effects model known as a random coefficients regression model for repeated measurement, will be conducted to evaluate and compare the rate and pattern of change over the 6 weeks in the MBSR and wait-listed control groups for pain catastrophizing.
Change in Mindfulness as measured by the Mindful Attention Awareness Scale | baseline, week 1, week 3, and week 6
  Descriptive statistics will be used to summarize mindfulness at week1, 3, and 6, as measured by the Mindful Attention Awareness Scale. Trajectory analyses, using a type of mixed effects model known as a random coefficients regression model for repeated measurement, will be conducted to evaluate and compare the rate and pattern of change over the 6 weeks in the MBSR and wait-listed control groups for pain catastrophizing.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Tanabe, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University School of Nursing, Durham, North Carolina, United States

REFERENCES:
- [Derived] Williams H, Silva S, Simmons LA, Tanabe P. A telephonic mindfulness-based intervention for persons with sickle cell disease: study protocol for a randomized controlled trial. Trials. 2017 May 15;18(1):218. doi: 10.1186/s13063-017-1948-x. PMID 28506281